CLINICAL TRIAL: NCT06350903
Title: Suppression With Empagliflozin as an Alternative To High-Fat Low-Carbohydrate Diet for Myocardial FDG-PET Imaging
Brief Title: Suppression With Empagliflozin as an Alternative To High-Fat Low-Carbohydrate Diet for Myocardial F-fluorodeoxyglucose Positron Emission Tomography (FDG-PET) Imaging
Acronym: SWEET-HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthieu Pelletier-Galarneau, MD MSc (Other)
Responsible Party: Sponsor-Investigator, Matthieu Pelletier-Galarneau, MD MSc, Chief, division of nuclear medicine at Institut de cardiologie de Montreal, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: ICM 2024-3356
Record Dates: First submitted 2024-03-18; First posted 2024-04-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2024-10

CONDITIONS: Myocardial Suppression
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fast + High-fat low-carbohydrate diet — Participants will be instructed to follow a strict HFLC diet starting on the morning of the day before the visit and to fast for 14 hours, starting at 7pm the day before the visit. Participants will be allowed to drink water and take their medications.
Combination Product: Fast + Empagliflozin — Participants will be instructed to fast for 14 hours, starting at 7pm the day before the visit. Participants will be allowed to drink water and take their medications. Participants will also be instructed to take an oral dose of 50 mg of empagliflozin at 7am the morning before the experimental visit and on the day of the experimental visit.

SUMMARY:
The overall objective of this study is to assess if the empagliflozin has the potential to substitute the high fat low carb (HFLC) diet for the preparation of cardiovascular FDG-PET studies.

DETAILED DESCRIPTION:
The overall objective of this study is to assess if the SGLT2 inhibitor empagliflozin has the potential to substitute the high fat low carb (HFLC) diet for the preparation of cardiovascular FDG-PET studies. This study will evaluate if an acute administration of empagliflozin (tablets of 10 and/or 25 mg) combined with fasting can sufficiently increase the BHB levels, a proxy of myocardial FDG uptake.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years
2. Ability to follow the HFLC diet
3. Ability to provide informed consent

Exclusion Criteria:

1. Treated with SGLT2 inhibitors
2. History of hypersensitivity or allergy to empagliflozin
3. Hypotension with blood pressure <100/65 mmHg
4. Strict vegan
5. Pregnancy
6. Breastfeeding
7. Type I or type II diabetes
8. Renal failure with Estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.72m2
9. Receiving steroids
10. History of diabetic ketoacidosis (DKA)
11. History of hypoglycemia
12. Any condition that, in the opinion of the investigator, could compromise the participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Levels of serum Beta-hydroxybutyrate (BHB) mmol/L | 1 day
  Average differences in serum levels of BHB measured following a fast and administration of empagliflozin versus following a fast preceded by a HFLC diet

SECONDARY OUTCOMES:
Proportions of serum Beta-hydroxybutyrate (BHB) >0.5 mmol/L | 1 day
  Proportion of participants with serum BHB >0.5 mmol/L following a fast and administration of empagliflozin versus following a fast preceded by a HFLC diet.
Proportions of glycemia levels (mmol/L) <3.5 mmol/L | 1 day
  Proportion of participants with glycemia <3.5 mmol/L following a fast and administration of empagliflozin versus following a fast preceded by a HFLC diet.
Acceptability and tolerance of each protocol, as reported by patients by a dedicated survey. | Through study completion, up to 3 months.
  Proportion of participants who preferred the empagliflozin to the HFLC diet as assessed by a dedicated survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided